CLINICAL TRIAL: NCT07160751
Title: Observation of Cognitive Complaints in Patients With Localized, Operable Non-small Cell Lung Cancer
Brief Title: Cognition and Patients With Lung Cancer
Acronym: COGNIPULM
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250754
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Localized, Operable Non-small Cell Lung Cancer
Keywords: localized; Operable non-small cell lung cancer,; Cognitive complaints
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgery only
  Interventions: Other: Self-questionnaire
- Neoadjuvant treatment (chemotherapy or chemoimmunotherapy) followed by surgery
  Interventions: Other: Cognitive tests
- Surgery followed by adjuvant treatment (chemotherapy)
  Interventions: Other: Assessment of the impact of social vulnerability on patient complaints

INTERVENTIONS:
Other: Self-questionnaire — FACT-Cog, HADS, FA12, EPICES, socio-professional and socio-demographic questionnaire
  Groups: Surgery only
Other: Cognitive tests — Hopkins Verbal Learning Test (HVLT). Trail Making Test (TMT). Verbal fluency test. Digit memory WAIS-IV.
  Groups: Neoadjuvant treatment (chemotherapy or chemoimmunotherapy) followed by surgery
Other: Assessment of the impact of social vulnerability on patient complaints — EPICES at month 12
  Groups: Surgery followed by adjuvant treatment (chemotherapy)

SUMMARY:
Cognitive complaints in patients treated for cancer can impact their quality of life.

Studies show that these cognitive complaints may have multifactorial origins and appear at different stages of the care pathway.

In a population of patients treated for confirmed localized non-small cell lung cancer (NSCLC), this study aims to detect and monitor the onset of cognitive complaints over time.

The timing of the complaints during the treatment, the cognitive functions affected (memory, attention, concentration…), as well as the perceived intensity of the discomfort, will be examined.

The study also explores the influence of co-factors such as mood, fatigue, socio-cultural status, and level of social vulnerability on these cognitive complaints.

DETAILED DESCRIPTION:
Chemofog" is the term used to describe cognitive difficulties associated with cancer treatments, such as chemotherapy, radiotherapy, and surgery.

These difficulties may include problems with memory, executive functions, attention, orientation, verbal comprehension, and information processing speed, and can occur during and after treatment.

Although generally mild to moderate, they can limit patients' ability to return to work and manage daily tasks. These cognitive difficulties are often associated with mood changes and increased fatigue.

They significantly impair functional independence and quality of life for cancer patients.

A baseline assessment of cognitive function prior to treatment is essential. Various factors-such as age, medical or psychiatric history, social vulnerability, or other neurological and psychological risk factors-may preexist the cancer diagnosis.

Subsequently, the impact of the disease itself, the treatments, changes in socio-professional status, and increased or induced socioeconomic hardship, as well as psychological upheaval (such as receiving the diagnosis, anxiety, or family disruptions), may all lead to cognitive disturbances.

These disturbances, referred to as Cancer-Related Cognitive Impairment (CRCI), affect the quality of life of cancer survivors.

According to one study, 26% of lung cancer survivors present with CRCI.

Biological and genetic factors such as cellular senescence, inflammatory processes, and DNA damage are thought to play a role in the development of CRCI.

Current research seeks to identify relevant biomarkers of cognitive decline, such as cytokine levels, to better understand its mechanisms and improve its management.

Various risk factors for CRCI have been identified: advanced age, lower baseline cognitive functioning, and lack of physical activity.

Cognitive complaints have been recognized for more than 20 years and may affect up to 75% of cancer patients, regardless of cancer type.

Yet too few patients are informed of the existence of CRCI, even though awareness of these issues can directly impact their abilities-particularly in the professional sphere.

A French-language framework and international guidelines have been developed to help standardize cognitive assessment.

Nevertheless, the absence of methodological consensus on the selection of variables (biomarkers, cognitive tests, adjustment factors), measurements, analysis of results, and timing of evaluations leads to these difficulties being underdiagnosed.

Thus, further studies are needed to investigate this subject and ultimately implement appropriate management strategies.

Based on the recommendations of the Association Francophone des Soins Oncologiques de Support (AFSOS), which emphasize the importance of raising clinicians' awareness of the "chemofog/CRCI" issue-both to better define cognitive complaints and to propose appropriate management-our study aims to examine cognitive complaints in individuals diagnosed with confirmed, operable, localized non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 to 74 years
* Suspected or confirmed localized and operable non-small cell lung cancer (NSCLC)
* Surgical treatment with or without perioperative systemic medical therapy
* Ability to independently complete self-questionnaires via the Cleanweb platform
* Patients with access to a phone, tablet, or computer at home to complete the electronic self-questionnaires.

Exclusion Criteria:

* Known pre-existing cognitive disorders
* Presence on the day of inclusion of one or more factors causing mental confusion: electrolyte imbalances, renal failure, hepatic failure, infections, bladder distension, fecal impaction
* Known psychiatric or neurological diseases (e.g., multiple sclerosis, Parkinson's disease, dementia, stroke, traumatic brain injury with loss of consciousness)
* Current use of neuroleptic treatments
* History of cancer treatment within the past 10 years
* Fibromyalgia
* Individuals who cannot read French or are not French-speaking
* Patients who have never attended school

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population includes adults aged 18 to 74 years with suspected localized and operable non-small cell lung cancer. Patients whose cancer diagnosis is not confirmed after inclusion will be prematurely withdrawn from the study
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
To examine the onset, intensity and duration of the PCI (Perceived Cognitive Impairment) score | 12 months
  Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) self-report questionnaire : min =0, max=132

SECONDARY OUTCOMES:
Determine whether there is a clinical and/or social phenotype associated with cognitive complaint. | 12 months
  Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) : min = 0, max=132
Determine whether there is a clinical and/or social phenotype associated with mood | 12 months
  Hospital Anxiety and Depression scale (HADS) : min=0, max=42
Determine whether there is a clinical and/or social phenotype associated with fatigue | 12 months
  European Organisation for Research and Treatment of Cancer - Fatigue Scale (EORTC QLQ-FA12) : min=0, max=100
Assessment of the impact of perioperative surgical and medical treatments on cognitive complaint | 12 months
  Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) : min=0, max=132
Assessment of the impact of perioperative surgical and medical treatments on mood. | 12 months
  Hospital Anxiety and Depression scale (HADS ): min=0, max=42
Assessment of the impact of perioperative surgical and medical treatments on fatigue. | 12 months
  European Organisation for Research and Treatment of Cancer - Fatigue Scale (EORTC QLQ-FA12) : min=0, max=100
Objective assessment via cognitive tests of the impact of cancer, treatments and co-factors on patients' cognition | 12 months
  Cognitive tests recommended by the International Cognition and Cancer Task Force (ICCTF) :
  Hopkins Verbal Learning Test (HVLT). Trail Making Test (TMT). Verbal fluency test. Digit memory WAIS-IV.
Assessment of the impact of social vulnerability on patient complaints | 12 months
  Assessment of Precarity and Health Inequalities in Health Examination Centers (EPICES): min = 0, max = 100.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle HARDY LEGER, Principal Investigator — Hôpital Cochin, Assistance Publique-Hôpitaux de Paris - Service de pneumologie.
Locations (1):
- Hôpital Cochin - Service de pneumologie, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No